CLINICAL TRIAL: NCT04301453
Title: The Effect of Maternal Scent on Sleep Wake States, Brain Maturation, and Heart Rate Variability: A Randomized Controlled Trial
Brief Title: The Effect of Maternal Scent on Sleep Wake States
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Columbia University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: AAAS5200
Record Dates: First submitted 2020-03-06; First posted 2020-03-10 (Actual); Last update posted 2022-08-26 (Actual); Status verified 2022-08

CONDITIONS: Development, Infant
Keywords: Sleep wake cycles; Quiet sleep; Active sleep; Maternal scent

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Maternal Scent Group (Experimental): Infants in this group will be exposed to a breast pad worn by their mothers to extract maternal scent. This exposure will last 24 hours.
  Interventions: Other: Maternal Scent
- Control Group (No Intervention): Infants in this group will receive standard of care.

INTERVENTIONS:
Other: Maternal Scent — Mothers will wear a breast pad during their visit. The breast pad will be placed in the hats of infants for 24 hours.
  Arms: Maternal Scent Group

SUMMARY:
This study will be a prospective, randomized controlled study, which aims to determine if a maternal scent intervention improves the sleep wake states, brain maturation, and heart rate variability in premature infants admitted to the neonatal intensive care unit (NICU). Infants will be randomized to either 24 hours of exposure to maternal scent or standard of care. Sleep wake states will be obtained using behavioral coding. Brain maturation will be measured using several electroencephalogram (EEG) parameters. Heart rate variability will be collected as part of vital sign collection.

DETAILED DESCRIPTION:
Sleep is important for the growth and development of infants. There are different states that make up sleep wake cycles including quiet sleep, active sleep, and transitional sleep. The amount of time that infants spend in quiet sleep increases as they mature. There are different tools that can be used to measure sleep state including EEG, behavior, and vital signs. Recent research has looked at ways to improve sleep in infants admitted to the NICU including music and maternal voice. The investigators are interested in studying maternal scent. Maternal scent has been shown to improve infant feeding and to reduce infant crying during painful procedures. Therefore, the investigators are interested in studying how maternal scent might affect sleep wake state in infants admitted to the NICU. The investigators will observe infant behavior and use EEG and vital signs to assess sleep state in infant after they are exposed to maternal scent.

ELIGIBILITY:
Inclusion criteria:

* Infants born at 30 weeks gestation to 36 weeks gestation.

Exclusion criteria:

* Infants with congenital anomalies, neonatal abstinence syndrome, or head ultrasound findings of grade II intraventricular hemorrhage or greater.
* Infants participating in studies with similar interventions.

Ages: 30 Weeks to 36 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 78 (Actual)
Dates: Start 2019-10-30 (Actual); Primary Completion 2021-05-27 (Actual); Study Completion 2021-05-27 (Actual)

PRIMARY OUTCOMES:
Percentage of time spent in quiet sleep | 2 hours
  Active sleep, quiet sleep, and indeterminate sleep will be behaviorally coded to determine the total amount of time spent in quiet sleep.
Percentage of time spent active sleep | 2 hours
  Active sleep, quiet sleep, and indeterminate sleep will be behaviorally coded to determine the total amount of time spent in active sleep.

SECONDARY OUTCOMES:
Beta to theta ratio | 2 hours
  EEG data will be analyzed to determine the beta to theta ratio in order to assess sleep wake cycling.
Number of mothers diagnosed with acute stress disorder based on score on the Stanford Acute Stress Reaction Questionnaire (SASRQ) | 2 hours
  The SASRQ questionnaire is used to assess symptoms of stress after a difficult event. There are four sub-scales including 1) Dissociative Symptoms 2) Re-Experiencing 3) Avoidance and 4) Increased Anxiety. These sub-scales are scored to determine if the diagnosis of acute stress disorder can be made. A symptom is scored as present if the respondent marks it as occurring at least "sometimes," which includes a response of 3, 4 or 5 on the 0-5 scale. A diagnosis of Acute Stress Disorder requires at least 3 symptoms out of the five types of dissociative symptoms, 1 reexperiencing symptom, 1 avoidance symptom, and 1 marked anxiety/increased arousal symptom. In order to count a symptom as present, circled response must be 3 or higher.

CONTACTS AND LOCATIONS:
Overall Officials: Rakesh Sahni, MD, Principal Investigator — Columbia University
Locations (1):
- New York Presbyterian, Columbia University Medical Center, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No